CLINICAL TRIAL: NCT02821598
Title: Effects of the Proprioceptive Neuromuscular Facilitation for Promoting Muscular Irradiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Aline de Souza Pagnussat, PhD, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 888.006
Record Dates: First submitted 2016-06-22; First posted 2016-07-01 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Motor Disorders
MeSH Terms: conditions — Motor Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (5):
- Upper limb pattern (Experimental): Upper Limb pattern with flexion - abduction - external rotation
  Interventions: Other: Upper Limb pattern with flexion - abduction - external rotation
- Lower limb pattern 1 (Experimental): Lower Limb pattern with flexion - adduction - external rotation with knee flexion;
  Interventions: Other: Lower Limb pattern with flexion - adduction - external rotation with knee flexion
- Lower limb pattern 2 (Experimental): Lower Limb pattern with flexion - abduction - internal rotation with knee flexion;
  Interventions: Other: Lower Limb pattern with flexion - abduction - internal rotation with knee flexion
- Lifting to the right (Experimental)
  Interventions: Other: Lifting to the right
- Sit to Stand (Active Comparator): Sit to Stand task
  Interventions: Other: Sit to Stand

INTERVENTIONS:
Other: Upper Limb pattern with flexion - abduction - external rotation — The PNF pattern will be applied three times. Participants will be in supine position under a stretcher, with arms folded and lower limbs in neutral position. In order to induce irradiation for the contralateral lower limb, the left foot sole will be kept in contact with the wall. For EMG recording, the participant will be positioned at the end of the PNF pattern and then the isometric contraction will be solicited. The command used was: "do not let me move you".
  Arms: Upper limb pattern
Other: Lower Limb pattern with flexion - adduction - external rotation with knee flexion — The PNF pattern will be applied three times. Participants will be in supine position under a stretcher, with arms folded and lower limbs in neutral position. In order to induce irradiation for the contralateral lower limb, the left foot sole will be kept in contact with the wall. For EMG recording, the participant will be positioned at the end of the PNF pattern and then the isometric contraction will be solicited. The command used was: "do not let me move you".
  Arms: Lower limb pattern 1
Other: Lower Limb pattern with flexion - abduction - internal rotation with knee flexion — The PNF pattern will be applied three times. Participants will be in supine position under a stretcher, with arms folded and lower limbs in neutral position. In order to induce irradiation for the contralateral lower limb, the left foot sole will be kept in contact with the wall. For EMG recording, the participant will be positioned at the end of the PNF pattern and then the isometric contraction will be solicited. The command used was: "do not let me move you".
  Arms: Lower limb pattern 2
Other: Lifting to the right — The PNF pattern will be applied three times. Participants will be in supine position under a stretcher, with arms folded and lower limbs in neutral position. In order to induce irradiation for the contralateral lower limb, the left foot sole will be kept in contact with the wall. For EMG recording, the participant will be positioned at the end of the PNF pattern and then the isometric contraction will be solicited. The command used was: "do not let me move you".
  Arms: Lifting to the right
Other: Sit to Stand — Subjects will be sitting on a chair without armrests with ankles positioned at approximately 10 degrees of dorsiflexion. Knees will be kept at approximately 100 degrees of flexion. During the task, the participant will be instructed to stand from the sitting position while keeping their arms crossed over the chest. The examiner will give the command "ready - set - go". The task will be performed three times.
  Arms: Sit to Stand

SUMMARY:
This study aims to evaluate the effects of Proprioceptive Neuromuscular Facilitation (PNF) patterns delivered to the upper limb, lower limb and trunk for promoting motor irradiation to the contralateral lower limb.

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* sedentary
* healthy
* body mass index between 18.5 - 24.9 kg/m2

Exclusion Criteria:

* having any injuries that prevented the implementation of the proposed activities
* being pregnant

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Muscular activity by means of Electromyography | Change from pre to post intervention (at least 40 min)
  Muscular activity will be assessed in the left lower limb

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil